CLINICAL TRIAL: NCT02493088
Title: Passage à l'Acte en Maison d'arrêt : Recherche d'éléments Contextuels récurrents Prospectifs et rétrospectifs
Brief Title: Conduct Disorder in Prison: Search for Prospective and Retrospective Recurring and Contextual Elements
Acronym: CoDiRCE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2014P08040
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Antisocial personality: Individuals Diagnosed with Antisocial Personality Disorder
  Interventions: Other: Antisocial personality recording of behavior and contextual elements

INTERVENTIONS:
Other: Antisocial personality recording of behavior and contextual elements — aberrant driving behaviors and upstream contextual elements of individuals diagnosed with antisocial personality disorder will be recorded during the study

SUMMARY:
The prediction of dangerousness remains a delicate subject, relevant in current psychiatry. Scalable psychopathological elements identified in schizophrenia and mood disorders are considered as most at risk for crime committing. The French High Authority of Health (HAS) recommends to identify and prevent risk situations of violence and to develop research at this level. Some authors have worked on criminal career and became interested in risk factors for aberrant driving behaviors but also in environmental or clinical elements accompanying these phases. To our knowledge, no specific study about contextual elements before misconduct and which could lead to aberrant driving behaviors among individuals diagnosed with antisocial personality disorder has been described to date The investigators propose to follow individuals diagnosed with antisocial personality disorder in prison during 6 months in order to list their conduct disorders and contextual elements upstream of these misconducts. The investigators will also study the effect of contextual factors related to judicial steps on the appearance of aberrant driving behaviors.

DETAILED DESCRIPTION:
This study aims at identifying elements that can provoke frustration and lead to aberrant driving behaviors. The question is whether there are triggers that occur more frequently for the same subject. If so, these specific contextual elements could be detected in order to prevent violent acts.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Over 18
* Detention sentence in prison in Rochefort between March and August 2015
* Positive psychopathy score at PCL-R (Psychopathy Checklist-revised) test: score greater than or equal to 30

Exclusion Criteria:

* Chronic psychosis
* Bipolar disorder
* Women
* Minors,
* negative score at the PCL-R
* Subject under protection measure (curator or guardian)
* Refusal to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with antisocial personality disorder have been chosen for this study due to their propensity of aberrant driving behaviors, including torts.
  Individuals detained in prison Rochefort and with a despcription fitting a psychopathic profile (impulsive, lack of empathy, repeated misconducts, repeat offenses ...) are informed of the study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PARRY, MD, Principal Investigator — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Maison d'arrêt de Rochefort, Rochefort, France

REFERENCES:
- [Background] Haute Autorité de Santé. Dangerosité psychiatrique : étude et évaluation des facteurs de risque de violence hétéro-agressive chez les personnes ayant des troubles schizophréniques ou des troubles de l'humeur. In: Service des bonnes pratiques professionnelles. Saint-Denis La Plaine: Service documentation - information des publics; 2011.
- [Background] Quinsey VL, Harris GT, Rice ME, Cormier CA. Violent Offenders: Appraising and Managing Risk, Second Edition. American Psychological Association. Washington, DC, US 2006. 462 p.
- [Background] Moulin V, Favard A-N.
- [Background] Moulin V, Senon J-L. Évaluation de la dynamique criminelle et des processus qui sous-tendent l'agir infractionnel dans un cadre expertal, 2010.
- [Background] Litinetskaia M. Dangerosité, délinquance et passage à l'acte : psychopathologie et prédictivité. Annales médico-psychologiques 170. 99-102; 2012.
- [Background] Côté G. Vers une définition de la psychopathie. Pham TH & Côté. Villeneuve d'Ascq, France: Presse Universitaire du Septentrion; 2000. 240 p.
- [Background] Balier C. Psychanalyse des comportements violents. Puf. Rouge LF. Paris1988
- [Background] Gravier B. Violence et psychopathie. Psychiatrie légale et criminologie clinique. Issy-les-Moulineaux : Elsevier Masson, 2013. Les âges de la vie. ISBN : 978-2-294-73163-1; 2013.
- [Background] Hare RD, Craigen D. Psychopathy and physiological activity in a mixed-motive game situation. Psychophysiology. 1974 Mar;11(2):197-206. doi: 10.1111/j.1469-8986.1974.tb00839.x. No abstract available. PMID 4821619
- [Background] Vanderstukken O. Troubles de l'attention et des fonctions executives chez les psychopathes. Université catholique de Louvain;1998.
- [Background] Pham TH. [Psychometric evaluation of the Hare Psychopathy Questionnaire in a Belgian prison population]. Encephale. 1998 Sep-Oct;24(5):435-41. French. PMID 9850817
- [Background] Etude de Cote G, Sheilagh H, Toupin J. citée par Pham TH, Cote G. Psychopathie : Théorie et Recherche. Septentrion Presse Universitaire; 2000.
- [Background] Sreenivasan S, Kirkish P, Eth S, Mintz J, Hwang S, Van Gorp W, Van Vort W. Predictors of recidivistic violence in criminally insane and civilly committed psychiatric inpatients. Int J Law Psychiatry. 1997 Spring;20(2):279-91. doi: 10.1016/s0160-2527(97)00008-3. No abstract available. PMID 9178068
- [Background] Méry B. Diplôme Inter-Universitaire de psychiatrie criminelle et médicolégale. "Organisation du système pénitentiaire " ; Mars 2014.
- [Background] Hare RD, Neumann CN. The PCL-R Assessment of Psychopathy: Development, Structural Properties, and New Directions. C. Patrick ed. New York: Guilford; 2006.
- [Background] Cote G, Hodgins S, Toupin J. Psychopathie : Prévalence et spécificité clinique. Psychopathie : théorie et recherche. Paris : Septentrion Presse Universitaire, 2000, p 47-75. ISBN 2-85939-612-8; 2000.
- [Background] COTE G., HODGINS S., TOUPIN J. Psychopathie : Prévalence et spécificité clinique. Psychopathie : théorie et recherche. Paris : Septentrion Presse Universitaire, 2000, p 47-75. ISBN 2-85939-612-8. 2000.
- [Background] Salekin RT, Rogers R, Sewell KW. Construct validity of psychopathy in a female offender sample: a multitrait-multimethod evaluation. J Abnorm Psychol. 1997 Nov;106(4):576-85. doi: 10.1037//0021-843x.106.4.576. PMID 9358688
- [Background] Ministère de la Justice, Statistiques trimestrielles de la population prise en charge en milieu fermé [Consulté le 30/01/2015]. Disponible à partir de l'URL : http://www.justice.gouv.fr/art_pix/trimestrielle_MF_janvier_2014.pdf - Tableau 1. 2014.)
- [Background] Pham TH. L'évaluation de la psychopathie. Psychiatrie légale et criminologie clinique. Les âges de la vie. Issy-les-Moulineaux : Elsevier Masson; 2000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 3 2015 to May 30 2015 Rochefort prison
Pre-assignment Details: Patient with a negative psychopathy score at PCL-R were excluded A patient was transfered before assignment
Period: Overall Study
Arm/Group | Antisocial Personality
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Antisocial Personality
Number analyzed (Participants) | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [18 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  France | 11

OUTCOME MEASURES:

1. Primary Outcome: The Number of Individuals Diagnosed With Antisocial Personality Disorder in Rochefort Prison With Aberrant Driving Behaviors.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Antisocial Personality
Number analyzed (Participants) | 11
participants | 9

2. Secondary Outcome: Percentage of Aberrant Driving Behaviors With Contextual Element Observed Before Aberrant Driving Behaviors
Description: Collected contextual elements were :
  * Disorders in the institution (with a caregiver, frustration with the rules)
  * Difficulty / frustration with an inmate
  * Difficulty / frustration with the entourage
  * Consumption of alcohol or other toxic substances
  * Steps in the judicial process (refusal of parole, reduction of sentence ...)
  * Psychiatric symptoms: delirious, sleep disorders, nightmares The numerator for the percentage calculated is the number of aberrant driving behaviors with contextual element.
  The denominator for the percentage calculated is the total number of aberrant driving behaviors (with and without contextual element)
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percent of aberrant driving behaviors
Units Other Than Participants: Number of aberrant driving behaviors
Arm/Group | Antisocial Personality
Number analyzed (Participants) | 11
Number analyzed (Number of aberrant driving behaviors) | 46
percent of aberrant driving behaviors | 67.4 [53.8 to 80.9]

3. Secondary Outcome: Number of Observed Situations Per Type of Aberrant Driving Behavior (Auto-aggressive, Aggressive or Other Hetero Transgression)
Description: Auto-aggressive: attempted suicide, any gesture of mutilation (scarification, punching in a wall, etc.) Aggressive: rixes with fellow inmates or prison staff, attempted homicides, sexual assaults, etc.
  Other hetero transgression: Failure to comply with the rules of the institution, illegal entry of illicit objects into the establishment, consumption of toxic materials, destruction of property, etc.
Time Frame: 6 months
Measure: Number; unit: number of observed situations
Arm/Group | Antisocial Personality
Number analyzed (Participants) | 11
number of observed situations
  auto-aggressive | 0
  aggressive | 15
  other hetero transgression | 31

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Antisocial Personality: Individuals Diagnosed with Antisocial Personality Disorder
  Aberrant driving behaviors and upstream contextual elements of individuals diagnosed with antisocial personality disorder were recorded during the study.
  Adverse events were not related to the study.
  Recorded adverse events were situations where subjects were harmed and required medical intervention.
Arm/Group | Antisocial Personality
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antisocial Personality (N=11)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1) — Lesions following a brawl with another inmate: cerebral contusion
Contusions (Injury, poisoning and procedural complications) | 1 (1) — Taken care in the emergency room after a fight with another co-detainee : multiple contusions due to punches Taken in the emergency room after a fight with another co-detainee: multiple contusions due to punches

LIMITATIONS AND CAVEATS:
data collected by healthcare workers (no 24/7 recording of behaviors). Too small sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes